CLINICAL TRIAL: NCT02666313
Title: WEB-Based Physiotherapy for People With Axial Spondyloarthritis: A Cohort Study
Brief Title: WEB-Based Physiotherapy for People With Axial Spondyloarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Lorna Paul (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Dr Lorna Paul, Reader in Rehabilitation, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEBPASS
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise — The physiotherapist will select exercises which are appropriate to that participant. Participants will complete online exercise diaries which are reviewed remotely by the physiotherapist. Depending on progress, exercises can be progressed, added or removed from the patient's individualised programme.
  Participants will be encouraged to undertake their exercise programme, according to evidence base guidelines, five days/week for 30 minutes/day. Participants will receive weekly phone calls for the first two weeks of the programme. Thereafter, every two weeks the physiotherapist will review the exercise diary of each participant and remotely alter the participant's exercise programme as appropriate, by changing any combination of exercises, level of difficulty or number of repetitions.

SUMMARY:
Regular exercise is a core component of the long-term management of people with axial spondyloarthritis (axial SpA). However, delivering long-term exercise programmes is unrealistic and unsustainable using traditional NHS services. Web-based physiotherapy, has been developed, a possible alternative service model to support people with axial SpA to exercise regularly however long-term compliance to the programme (12 months) needs to be established. The aim of this prospective cohort study is to assess the feasibility, sustainability and acceptability of a 12 month individualised web-based physiotherapy programme in people with axial SpA. Fifty people with established axial SpA, will receive 12 months of individualised, remotely monitored, web-based physiotherapy. The primary outcome will be four weekly compliance rates with the programme over the 12 month period. Secondary outcomes (baseline, 6 and 12 months) will include function, disease activity, spinal mobility, quality of life, attitudes and motivations towards exercise, fitness, health status, employment, physical activity. The number of interactions with health care professionals and changes in medication will be documented. A subsample of the cohort will be interviewed at 6 and 12 months to gather participants' views of the web-based physiotherapy programme and factors influencing compliance with the programme.

DETAILED DESCRIPTION:
Background and Rationale Axial spondyloarthritis (axial SpA) is an inflammatory arthritis characterised by inflammatory back pain and includes both ankylosing spondylitis (AS) and non-radiographic axial SpA. Axial SpA is associated with pain and stiffness in the spine and/or sacroiliac joints, reduced spinal mobility, fatigue, reduced physical activity, psychological consequences such as depression, and reduced function, work productivity and quality of life. Effective management in axial SpA requires a combination of pharmacological and non-pharmacological interventions. While there have been significant advances in pharmacological therapies, particularly with the introduction of TNF-inhibitors, there have been few advances in how physiotherapy and the non-pharmacological therapies are delivered. This is despite physiotherapy being recognised as the 'cornerstone' in the overall management of people with AS, in terms of both managing symptoms and maintaining function. Physiotherapy comprises of education and exercise programmes aimed at improving or maintaining spinal mobility, reducing spinal pain, increasing strength and stabilising or slowing down disability progression. Physiotherapy is required long-term and in combination with pharmacological therapies. A Cochrane Review in 2008 concluded that both home and supervised individual exercises were beneficial for people with AS, with group exercise more beneficial than home-based exercise. However, to be beneficial, exercise needs to be done at least five times per week, for at least 30 minutes per session and continued on a long-term basis. Patients with axial SpA are increasingly diagnosed and treated earlier, have reduced disease activity as a result of treatment with TNF-inhibitors and are more likely to be younger and in employment than was traditionally the case. For these reasons, patients find it difficult to attend and maintain regular traditional physiotherapy sessions, particularly in the long-term. Practically, then, exercise programmes must include some degree of home-based exercise since this level of exercise cannot be delivered on a long-term basis by the NHS or other services. Despite the requirement for regular physiotherapy, a recent NASS patient survey revealed that 60% of patients had not had physiotherapy in the previous 12 month period. There is therefore a need to find alternative service models which support and facilitate people with axial SpA to exercise regularly and on a long-term basis.

The Office of National Statistics reported that 86% of the adult population (aged over 16 years) in the UK had used the internet and 73% (36 million adults) used it on a daily basis. In addition, there are increasing numbers of people using the internet for health care information and resources. Thus the almost ubiquitous availability and use of the internet provides an ideal opportunity to deliver tailored, individualised, interactive exercise programmes for people with long-term conditions, including axial SpA. Web-based interventions are available 24 hours a day and thus the patient can choose the time and location in which they participate to suit their own personal circumstances. Physiotherapy-led, personalised web-based exercise therefore offers a potentially cost-effective mechanism to deliver this important long-term component in axial SpA and warrants evaluation.

Two groups based in the Netherlands have examined web-based interventions to increase physical activity in patients with rheumatoid arthritis (RA) and osteoarthritis (OA). Van Den Berg compared a 12 month individually targeted, physical intervention delivered online with 12 months of general online advice and education regarding physical activity in people with RA. In addition, the intervention group received regular emails from the physiotherapist and also attended group meetings every 3 months. The study demonstrated that the intervention was effective in increasing the proportion of participants achieving the national physical activity recommendations compared to the general training group. There was no difference however in function or quality of life and the authors noted that the website usage reduced over time. The study by Bossen et al (2013) investigated an internet delivered physical activity programme but in patients with hip and/or knee OA. The Join2move programme was a nine-week programme of nine modules to be completed by the participant. The results showed an increase in physical activity and time spent in moderate intensity physical activity but not significantly more so than a waiting list control. The study reported high attrition rates which were attributed mainly to the fully automated nature of the intervention and absence of human contact or support. Thus there is some evidence for the use of web-based interventions to increase physical activity in people with RA or OA however no previous studies have investigated axial SpA nor regular physiotherapy delivered via the internet.

We have developed a website in collaboration with patient groups and the Scottish Accessible Information Forum which is a platform for delivering individualised web-based physiotherapy (demonstration page: www.webbasedphysio.com (log in: testphysiopatient@gmail.com, password: password). We have evaluated the short term effectiveness of this approach (maximum of 12 weeks) in a number of patient groups. Kelders et al. (2012) reported that not all users continue to use web-based interventions in the desired way and that as usage reduces so does the effectiveness of the intervention. Since the evidence base suggests that people with axial SpA should exercise five days per week, it is important to evaluate the compliance/adherence to this web-based physiotherapy programme over a longer period.

Study Design Pilot cohort study

Aim The aim of this prospective cohort study is to assess the feasibility, sustainability and acceptability of a 12 month individualised web-based physiotherapy programme in people with axial SpA.

Research objectives

* Over a one year period how often do people with axial SpA use the web-based physiotherapy programme?
* What do people with axial SpA think of the web-based physiotherapy programme?
* What can we do to help people with axial SpA use the web-based physiotherapy programme long-term?
* What is the effect of one year of web-based physiotherapy on pain, stiffness, physical function, physical activity, quality of life and employment?
* Which patients are most likely to benefit from the web-based physiotherapy programme?

Research questions Primary Research Questions

• What are the four weekly compliance rates with this web-based physiotherapy programme over a one year period?

Secondary Research Questions

* What are the views of users of this web-based physiotherapy programme?
* Why do people stop using this web-based physiotherapy programme?
* Is there an association between compliance and patient outcomes?
* What are the associations between baseline characteristics and compliance and/or patient outcomes?
* Which patients are most likely to benefit from the intervention?
* Does 12 months of web-based physiotherapy have the potential to positively alter pain, disease activity, functional ability, exercise capacity, quality of life, physical activity and employment in axial SpA?

Plan of Investigation Fifty people with confirmed axial SpA, will receive 12 months of individualised, remotely monitored, web-based physiotherapy. They will be asked to do their exercise programme five times per week. The main outcome will be compliance to the programme measured every four weeks. Secondary outcomes (baseline, 6 and 12 months) are function, disease activity, spinal mobility, quality of life, exercise capacity, health status, employment, physical activity, and attitude and motivations toward exercise. Interactions with health care professionals and medication usage will be documented using a weekly paper diary. A smaller sample of 10 participants, a mixture of participants who do and do not adhere to their programme (a maximum variation sample), will be interviewed at 6 and 12 months to gather their views of the web-based physiotherapy programme and factors affecting compliance.

Website development The website consists of a home page, exercise pages, exercise diary and an advice/information section. Each exercise page within the website consists of a video demonstrating the exercise, text explaining the exercise, an audio description of the exercise and a timer. The site contains a catalogue of exercises, each with four levels of difficulty, as well as a warm up and cool down. The website can be easily accessed via a personal computer, tablet or smart television and will is customised for use for patients with axial SpA.

The programme incorporates a number of behavioural change techniques known to be successful in promoting and maintaining exercise behaviour eg. goal setting and monitoring. We have mapped the behavioural change techniques within the current website with the Behaviour Change Techniques Taxonomy proposed by Michie et al. (2013). Currently the programme incorporates goals and planning, feedback and monitoring, shaping knowledge, natural consequences, comparison of behaviours, repetition and substitution and antecedents. The website is being continually revised and the functionality will be improved depending on the results of our other studies and also from the results of this mapping exercise. The current exercise catalogue has been adapted and expanded to include AS-specific exercises based on the popular Back to Action programme (http://nass.co.uk/back-to-action) produced by the National Ankylosing Spondylitis Society (NASS) (permission has already been granted by NASS) and specifically developed for patients with axial SpA. The NASS Back to Action programme is currently available as a pdf/app, so the proposed web-based physiotherapy programme differs in that it will be (a) individualised (b) based on effective behavioural change techniques (discussed above) and (c) interactive, being regularly monitored and altered remotely by the physiotherapist.

Study sites NHS Greater Glasgow and Clyde Health Board (Stobhill hospital, Gartnavel General, Glasgow Royal Infirmary, Southern General Hospital, Inverclyde Royal Hospital, New Victoria Hospital, Royal Alexandra Hospital).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of axial SpA (made by a Rheumatology consultant and fulfilling the ASAS criteria) (Rudwaleit et al. 2009)
* Under the care of a Rheumatology consultant in NHS Greater Glasgow and Clyde
* Minimum of 1 year since diagnosis
* Access to a personal computer/tablet or smart television with an email address and internet connection
* Over 18 years old
* A good understanding of English language

Exclusion Criteria:

* • Have had joint replacement surgery or spinal surgery within the last 6 months

  * Other significant co-morbidity which would preclude taking part in a regular exercise programme
  * Currently taking part in regular exercise (three times per week or more) and/or a regular physiotherapy programme
  * Currently participating in another clinical trial (rehabilitation or pharmacological)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of exercise sessions completed | One year
  based on the number of times the participants complete their exercise diary each week; as recorded on the website. The physiotherapist will record the number of completed exercise sessions each week and, from this, the mean number of sessions completed every four weeks will be calculated. Compliance will be analysed for each four-week period and for each 3-month period.

SECONDARY OUTCOMES:
Functional Ability | One year
  Using the Bath ankylosing spondylitis index (BASFI) a validated self-reported 10 item questionnaire evaluating the ability to function and cope with activities of daily living over the past week. Each question is scored on a 100mm visual analogue scale from no limitations (0 mm) to very severe functional limitation (100 mm). Lower scores indicate better function, while higher scores indicate more functional disability. The Minimum Clinically Important Difference (MCID), which is the minimum level of change of an outcome measure that is considered to be clinically relevant, for BASFI is 7mm (Calin et al. 1994).
Level of Physical Activity | One year
  will be objectively measured for one week using an activPAL activity monitor. The device is attached to the participant's thigh using a waterproof dressing and is worn continuously during the monitoring period, including during bathing/showering and swimming. Participants will also be asked to keep an activity diary during this period. The device categorises the posture as either sedentary (seated or lying), standing or walking. In addition the number of steps per day is recorded (Grant et al., 2006). The activPAL will be fitted to the participant at each assessment and will be instructed to remove the device after one week and post it back to the research team in a stamped addressed envelope provided to them. We have used this method of returning the device in other studies to good effect.
Disease Activity | One Year
  Measured through the Bath Ankylosing spondylitis disease activity index, (BASDAI) which is a validated self-reported 6 item questionnaire measuring disease activity on a 100mm visual analogue scale, from none (0 mm) to very severe (100 mm). Items included in the BASDAI are severity of fatigue, spinal and peripheral joint pain, localised tenderness and morning stiffness over the past week. Lower scores indicate lower disease activity. The MCID for BASDAI is 10mm (scale 0-100mm) (Garrett et al. 1994).
Spinal Mobility | One year
  Measured through the Bath Ankylosing Spondylitis Metrology Index (BASMI), which comprises five clinical measurements of the posture and movement of the spine and provides a score out of 10 of the participant's limitation of movement due to their AS (Jenkinson et al. 1994).
Employment and Productivity | One year
  Assessed through the Work, Productivity and Activity Impairment (WPAI) questionnaire which is a validated 18 item, disease specific, self-reported measure of quality of life
Health Status | One year
  Health status will be measured using the EQ-5D which is a performance measure of functional exercise capacity and involves the measurement of the distance an individual is able to walk for a total of six minutes on a hard, flat surface (Balke, 1963). The participant is instructed to walk at a comfortable pace and to take rests as required. The 6MWT will be undertaken following the established protocol and the distance walked during the six minutes will be recorded. Although not specifically validated in axial SpA it is a well recognised outcome measure in a range of chronic conditions including OA
Attitude to exercise | one year
  Attitude to exercise will be measured using the Exercise Attitude Questionnaire-18 which is a means of evaluating participants' attitudes towards exercise. It has 18 questions which are scored by the participant. The EAQ will allow us to study how a participants' attitude affects their compliance. Participants may complete this independently, those who encounter reading/writing problems may be assisted by the assessor, however they will be unable to influence scores through discussion of question interpretation.
Personal motivation to exercise. | One year
  Personal motivation to exercise will be measured using the Exercise Motivations Inventory -2 (EMI-2). It is a 51-item, multidimensional instrument designed to test theoretically derived predictions concerning the influences of personal exercise participation. The principle components are stress management, weight management, recreation, social recognition, enjoyment, appearance, personal development, affliction, ill-health avoidance, competition and fitness and health pressures. Each question is rated on a scale of 0-5. Participants' may complete this independently, those who encounter reading/writing problems may be assisted by the assessor, however they will be unable to influence scores through discussion of question interpretation.
Number of Interactions with Health professionals | over one year
  the number of interactions with health care professionals such as GP visits will be documented throughout the study and any changes to medication noted.
Participant views on the website | One year
  Telephone interviews will be undertaken with 10 participants at 6 and 12 month assessments. A sample of maximum variation will be taken for these interviews, based on the compliance rates. The interviews will gather participants' views of the web-based physiotherapy programme in relation to factors affecting compliance with the intervention. The interviews will explore issues directly related to the programme itself such as ease of use, content, difficulties experienced and the amount/content of contact with the therapist. Interviews will also explore other barriers to compliance and possible solutions identified by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PHD, Study Chair — University of Glasgow; Stefan Siebert, MD, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paul L, Coulter EH, Cameron S, McDonald MT, Brandon M, Cook D, McConnachie A, Siebert S. Web-based physiotherapy for people with axial spondyloarthritis (WEBPASS) - a study protocol. BMC Musculoskelet Disord. 2016 Aug 24;17(1):360. doi: 10.1186/s12891-016-1218-1. PMID 27553492